CLINICAL TRIAL: NCT06478082
Title: Virtual Reality Gaming to Improve Upper Limb Functionality in Children With Cerebral Palsy
Brief Title: Home-based Virtual Reality Rehabilitation for Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 885
Record Dates: First submitted 2024-03-06; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Cerebral Palsy
Keywords: Home-based rehabilitation; Virtual Reality; Upper limb
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with unilateral Cerebral Palsy (Experimental): All children have unilateral cerebral palsy and are between 1-18 years old
  Interventions: Device: Home-based virtual reality training

INTERVENTIONS:
Device: Home-based virtual reality training — 8-week training with an advised frequency of 30 minutes per day, for 5 days per week.

SUMMARY:
Rationale: In a way, VR-based gaming shows some similarities to Constraint-induced movement therapy. VR games are controlled unimanually or bimanually. When unimanually-controlled games are performed with the affected upper limb, movements of the unaffected hand are completely ineffective. This mimics the principle of forced use. To some degree, also bimanually-controlled games result in a forced use of the affected upper limb.

Additionally, VR could help in the engagement in rehabilitation programs, as virtual environments and gaming increases enjoyment and motivation, and therefore therapy adherence. Accordingly, VR-based gaming may have the potential to improve upper limb functionality in children with CP.

Objective: This study aims to investigate the feasibility of a home-based VR intervention to improve upper limb functionality in children with CP. Sub-objective: The validation of a self-developed upper limb assessment (Upper Limb Reaching Test).

Study population: Children and adolescents with unilateral CP (age 10-18 years old). Intervention: The intervention consists of VR-based rehabilitation with the Oculus Quest device. The training frequency and duration represents 2x15 minutes a day, five days a week, for a total of eight weeks. Therefore, this rehabilitation intervention should represent a total amount of 20 hours of rehabilitation. However, the total dosage is variable as the intervention is self-managed.

Main study parameters/endpoints: Logbook, System Usability Scale, Melbourne Assessment 2, Wall Arm Reaching Test, Elbow and shoulder range of motion.

ELIGIBILITY:
Inclusion Criteria:

* CP children with a unilateral or severely asymmetric, bilateral spastic movement impairment.
* Age 10-18 years old.
* Manual Ability Classification System (MACS) scores I, II or III.
* House classification of 1, 2 or 3.

Exclusion Criteria:

* Significant (persisting) motion sickness, or any other related adverse event in VR.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
Logbook | During the 8-week intervention period
  Participants keep a logbook in which they log the date of training, games played, duration of activity and enjoyment of game
System Usability Scale | After the 8-week intervention
  This questionnaire consists of 10 items regarding the usability of the virtual reality training. Scores ranging between 0-100, with a higher score indicating better usability

SECONDARY OUTCOMES:
Melbourne Assessment 2 | Before and after 8-week intervention
  Item 1,2,10 and 13 were measured to evaluate quality of upper limb movements, specifically reaching movements. Scores ranging between 0-33, with a higher score indicating better arm function.
Wall Arm Reaching Test | Before and after 8-week intervention
  A test to evaluate the reaching ability in children with cerebral palsy. Children have to alternate with their arm between the hip and a target on the wall as fast a possible in 30 seconds. Scoring starts at 0 and has no maximum. A higher score, indicates a better arm functioning.
Range of motion Elbow | Before and after 8-week intervention
  Passive and active range of motion of the extension of the elbow. Ranging between 0-180 degrees. Closer to 0 indicating better extension.
Rang om motion Shoulder | Before and after 8-week intervention
  Passive and active range of motion of the anteflexion of the shoulder. Ranging between 0-180 degrees. Closer to 180 indicating better anteflexion.

CONTACTS AND LOCATIONS:
Overall Officials: Noël Keijsers, Prof., Principal Investigator — Donders Institute for Brain, Cognition and Behavior, Radboud University
Locations (1):
- Sint Maartenskliniek, Ubbergen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No